CLINICAL TRIAL: NCT03527693
Title: Retrospective Observational Study on the Treatment of Knee Chondral Lesions in Arthroscopy With Autologous and Micro-fragmented Adipose Tissue
Brief Title: Micro-fragmented Adipose Tissue Injection Associated With Arthroscopic Procedures in Patients With Knee Osteoarthritis
Acronym: LOOK
Status: Completed | Type: Observational
Sponsor: Spotorno Foundation (Other)
Responsible Party: Principal Investigator, Gabriele Cattaneo, Doctor, Spotorno Foundation
Other Study IDs: protocol n° 164REG2016
Record Dates: First submitted 2018-04-27; First posted 2018-05-17 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Symptomatic Knee Osteoarthritis
Keywords: Knee Chondropathy, Osteoarthritis, Micro-fragmented fat.
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Lipogems injection — Micro-fragmented adipose tissue (10 cc) was injected intra-articular after the arthroscopic procedure (shaving or shaving + meniscectomy).

SUMMARY:
The study aims to evaluate the effects of a single intra-articular injection of micro-fragmented adipose tissue obtained with the Lipogems® system in patients affected by knee chondropathy. End-points were determined by evaluating the patients in terms of improvement in symptoms, functional recovery and radiographic appearance compared to baseline.

DETAILED DESCRIPTION:
Background: The social impact of degenerative diseases is steadily increasing, because of the continued rise in the mean age of the active population. Articular cartilage lesions are generally associated with disability and symptoms such as joint pain and reduced function, and remain a challenge for the orthopaedic surgeon. Several non-invasive solution have been proposed, but the results achieved to date are far from being completely satisfactory. Recently, new therapeutic approaches, such as the use of mesenchymal stem cells, have been developed. Among the many sources, the adipose tissue is nowadays considered one of the smartest, due to its abundance and easy access.

The aim of this retrospective study is to explore whether patients affected by symptomatic knee osteoarthritis treated with micro-fragmented adipose tissue associated with a chondral shaving procedure experience an improvement in symptoms and function.

Methods: Thirty-eight consecutive patients affected by symptomatic knee osteoarthritis were treated in 2015 with an arthroscopic procedure associated with an injection of autologous and micro-fragmented adipose tissue. Micro-fragmented adipose tissue was obtained using a minimal manipulation technique in a closed system. Clinical outcomes were determined at 1, 3, 6, and 12 months follow-up using Knee Injury and Osteoarthritis Outcome Score questionnaire and direct physical examination. Safety of the procedure, recording type and incidence of any adverse event, was also assessed.

ELIGIBILITY:
Inclusion Criteria:

* knee chondropathy grade > II (ICRS classification),
* constant pain and failure of conservative treatments (physiokinesitherapy, corticosteroids, HA and/or PRP) for at least 12 months.

Exclusion Criteria:

* immune-mediated (non-infectious) synovitis
* OA Kellgren-Lawrence grade >3
* axial defects >10°
* metabolic disorders
* BMI > 40

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is composed of consecutive patients affected by symptomatic knee chondropathy observed at the Orthopedic Unit of Santa Corona Hospital / Spotorno Foundation Pietra Ligure (SV) and all treated with Lipogems® between 01 January 2015 and 31 December 2015.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical improvement documented with KOOS (Knee Injury and Osteoarthritis Outcome Score). | 12 months
  Change in one or more of the 5 KOOS sub-scales (worst 0 - best 100) from baseline evaluation to 12 months follow-up. A minimum of 10 points improvement is considered a clinically relevant change.

SECONDARY OUTCOMES:
Incidence of treatment-related adverse events (AE) | 12 months
  Safety of the procedure, documenting characteristics and incidence of AE.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Cattaneo, MD, Principal Investigator — Spotorno Foundation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cattaneo G, De Caro A, Napoli F, Chiapale D, Trada P, Camera A. Micro-fragmented adipose tissue injection associated with arthroscopic procedures in patients with symptomatic knee osteoarthritis. BMC Musculoskelet Disord. 2018 May 30;19(1):176. doi: 10.1186/s12891-018-2105-8. PMID 29848328